CLINICAL TRIAL: NCT04414618
Title: Opaganib, a Sphingosine Kinase-2 (SK2) Inhibitor in COVID-19 Pneumonia: a Randomized, Double-blind, Placebo-Controlled Phase 2a Study, in Adult Subjects Hospitalized With SARS-CoV-2 Positive Pneumonia
Brief Title: A Study of Opaganib in Coronavirus Disease 2019 Pneumonia
Acronym: COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABC-110
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- opaganib (Active Comparator): Study participants will receive opaganib 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours
  Interventions: Drug: Opaganib
- placebo (Placebo Comparator): Study participants will receive placebo 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Opaganib — Study participants received opaganib 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours (pharmacological and/or supportive).
  Other Names: Yeliva; ABC294640
  Arms: opaganib
Drug: Placebo — Study participants received placebo 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours (pharmacological and/or supportive).
  Arms: placebo

SUMMARY:
This proof of concept study will take place in the US and other countries in approximately 15 clinical sites and will enroll about 40 hospitalized patients diagnosed with COVID-19 infection who have developed pneumonia and require supplemental oxygen. 20 patients will receive opaganib in addition to standard of care twice each day for 14 days. 20 will receive matching placebo in addition to standard of care unless the patient has been discharged from the hospital without requiring supplemental oxygen, in which case study drug will only be administered for 10 days. All participants will be followed up for 4 weeks after their last dose of study drug.

DETAILED DESCRIPTION:
Opaganib, a sphingosine kinase-2 (SphK2) inhibitor, has been broadly tested in Phase I/II studies. Extensive nonclinical data indicates both anti-viral and anti-inflammatory activity via selective SphK2 inhibition which may prove beneficial for treating COVID-19 infection and resulting pneumonia. This proof of concept study will take place in the US and other countries and will enroll about 40 hospitalized patients diagnosed with COVID-19 infection who have developed pneumonia and require supplemental oxygen. Half of the patients, i.e. 20 patients, will receive opaganib in addition to standard of care for 14 days. The other 20 will receive matching placebo (capsules that do not contain the medication) in addition to standard of care. Study drug will be administered every day for 14 days, twice each day, unless the patient has been discharged from the hospital without requiring supplemental oxygen, in which case study drug will only be administered for 10 days. All participants will be followed up for 4 weeks after their last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female ≥18 to ≤80 years of age
2. Proven COVID-19 infection per RT-PCR assay of a pharyngeal sample (nasopharyngeal or oropharyngeal) AND pneumonia defined as radiographic opacities on chest X-ray
3. The patient requires supplemental oxygen at baseline
4. The patient, guardian or legal representative has signed a written IRB-approved informed consent.

5) Male participants with female partners of child-bearing potential agree to one of the following methods of contraception during the treatment period and for at least 1 month after the last dose of study drug:

* Abstinence from penile-vaginal intercourse and agree to remain abstinent.
* Male condom, with female partner using a highly effective contraceptive method. (For further details regarding highly effective contraceptive methods please see section 9.3.)

In addition, male participants must refrain from donating sperm for the duration of the study and for 1 months after last dose of study drug.

Male participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration for at least 1 months after the last dose of study drug

Female participants:

A female participant is eligible to participate if she is:

1. not pregnant
2. not breastfeeding
3. not a woman of child-bearing potential (WOCBP, as defined in Section 9.3)
4. a WOCBP who agrees to use a highly effective method of contraception consistently and correctly during the treatment period and for at least 1 months after the last dose of study drug (please see further details on Section 9.3).

Exclusion Criteria:

1. Any co-morbidity that may add risk to the treatment in the judgement of the investigator.
2. Requiring intubation and mechanical ventilation
3. Patient having a do not intubate or do not resuscitate order
4. Oxygen saturation >95% on room air
5. Any preexisting respiratory condition that requires intermittent or continuous ambulatory oxygen prior to hospitalization
6. Patient is, in the investigator's clinical judgment, unlikely to survive >72 hours
7. Pregnant or nursing women
8. Unwillingness or inability to comply with procedures required in this protocol.
9. Corrected QT (QTc) interval on electrocardiogram (ECG) >470 ms for females or >450 ms for males, calculated using Friedericia's formula (QTcF)
10. AST (SGOT) or ALT (SGPT) > 2.5 x upper limit of normal (ULN)
11. Bilirubin >2.0 x ULN (except where bilirubin increase is due to Gilbert's Syndrome)
12. Serum creatinine >2.0 X ULN
13. Absolute neutrophil count <1000 cells/mm3
14. Platelet count <75,000/mm3
15. Hemoglobin <8.0 g/dL
16. Currently taking medications that are sensitive CYP3A4, CYP1A2, CYP2C9, or CYP2C19 or CYP2D6 substrates and have a narrow therapeutic index. These should be decided in discussion with the Medical Monitor on a case-by-case basis.
17. Currently taking medications that are strong inducers or inhibitors of CYP2D6 and CYP3A4. These should be decided in discussion with the Medical Monitor on a case-by-case basis.
18. Currently taking warfarin, apixaban, argatroban or rivaroxaban.
19. Current drug or alcohol abuse.
20. Currently participating in a clinical study assessing pharmacological treatments, including anti-viral studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Levitt, MD, PhD, Study Director — RedHill Biopharma Limited
Locations (9):
- United States (8):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Miami Cancer Institute, Miami, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Albany Medical Center, Albany, New York
  - Oregon Health & Science University, Portland, Oregon
  - Memorial Herman Southeast Hospital, Houston, Texas
  - Memorial Hermann, Memorial City Medical Center, Houston, Texas
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Opaganib: Study participants will receive opaganib 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours
  Opaganib: Study participants will receive either opaganib 2 x 250 mg capsules (500 mg) every 12 hours, in addition to standard of care (pharmacological and/or supportive).
- Placebo: Study participants will receive placebo 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours
  Placebo: Study participants will receive placebo 2 x 250 mg capsules (500 mg) every 12 hours, in addition to standard of care (pharmacological and/or supportive).
Period: Overall Study
Arm/Group | Opaganib | Placebo
Started | 23 | 19
Completed | 15 | 12
Not Completed | 8 | 7
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opaganib | Placebo | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Customized [Count of Participants; unit: Participants]
  <70 years | 20 | 15 | 35
  >=70 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 16 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Measurement of the Change in Oxygen Requirement From Baseline
Description: Maximal oxygen flow (L/min) was recorded daily for the 14 days of treatment for each participant. Participant individual area under the curve (AUC) was calculated based on the trapezoidal rule, after subtracting the baseline oxygen requirement at each day. The median AUC absolute change from baseline (L/min) for each treatment arm is presented.
Time Frame: 14 days
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication).
Measure: Median (95% Confidence Interval); unit: L/min*day
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
L/min*day | -38.8 [-56.5 to 0] | -33.0 [-149.5 to -12.5]

2. Secondary Outcome: Measurement of Time to the Reduction in Oxygen Requirement.
Description: The time required between arms to achieve 50% reduction from baseline in supplemental oxygen based on oxygen flow in L/min.
Time Frame: 14 days
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication). However, one subject who did not have supplemental oxygen requirement at randomization was excluded from this analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 21 | 18
Days | 5.00 [4.00 to 12.00] | 8.00 [4.00 to NA] — Some subjects didn't reach 50% reduction in oxygen requirement.

3. Secondary Outcome: The Percentage of Subjects no Longer Receiving Supplemental Oxygen for at Least 24 Hours by Day 14
Description: The percentage of subjects in each arm no longer requiring supplemental oxygen for at least 24 hours by Day 14.
Time Frame: 14 days
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
Participants | 11 | 4

4. Secondary Outcome: Time to Negative Swabs for SARS-CoV-2 by PCR Post Treatment
Description: The time in each arm to two consecutive negative swabs for SARS-CoV-2 by PCR nasopharyngeal or oropharyngeal swab, at least 24 hrs. apart.
Time Frame: 6 weeks
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication). However, as most subjects had been discharged by Day 7 and as the study was not designed to be performed on an outpatient basis, data was not available from enough subjects to perform these analyses.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
Days | NA [NA to NA] — As most subjects had been discharged by Day 7 and as the study was not designed to be performed on an outpatient basis, data was not available from enough subjects to perform these analyses. | NA [NA to NA] — As most subjects had been discharged by Day 7 and as the study was not designed to be performed on an outpatient basis, data was not available from enough subjects to perform these analyses.

5. Secondary Outcome: The Percentage of Subjects With at Least Two Consecutive Negative Swabs for SARS-CoV-2 by PCR at Day 14
Description: The percentage of subjects in each arm to achieve two consecutive negative PCR nasopharyngeal or oropharyngeal swabs for SARS-CoV-2 at Day 14, at least 24 hrs. apart.
Time Frame: 14 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Study participants received opaganib 2 x 250 mg capsules (500 mg) plus standard of care every 12 hours (pharmacological and/or supportive).
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
Participants | NA — As most subjects had been discharged by Day 7 and as the study was not designed to be performed on an outpatient basis, data was not available from enough subjects to perform these analyses. | NA — As most subjects had been discharged by Day 7 and as the study was not designed to be performed on an outpatient basis, data was not available from enough subjects to perform these analyses.

6. Secondary Outcome: Intubation and Mechanical Ventilation Requirements
Description: The percentage of patients in each arm who require intubation and mechanical ventilation by Day 14
Time Frame: From screening phase and every day from day 1 to day 14 of treatment
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
Participants | 2 | 2

7. Secondary Outcome: Evaluation of the Time to Intubation and Mechanical Ventilation
Description: The time in each arm for the patient to require mechanical ventilation.
Time Frame: From screening phase and every day from day 1 to day 14 of treatment
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
Days | NA [NA to NA] — The median time to intubation and mechanical ventilation was not reached in either group. | NA [NA to NA] — The median time to intubation and mechanical intubation was not reached in either group.

8. Secondary Outcome: Evaluation the Proportion of Patients, With at Least One Measurement of Fever at Baseline Who Are Afebrile at Day 14
Description: The proportion of patients in each arm, with at least one measurement of fever at baseline (defined as temperature >38.0 C[100.4 F]), who are afebrile (defined as temperature <37.2C [99 F]) at Day 14
Time Frame: From screening phase and every day from day 1 to day 14 of treatment
Population: Patients in the Modified ITT (mITT) population (randomized and treated with at least one dose of study medication) with at least one measurement of fever at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 3 | 0

9. Secondary Outcome: Evaluation of Mortality 30 Days Post-baseline
Description: The mortality in each arm 30 days post-baseline.
Time Frame: 30 days after day 1 of treatment
Population: Modified ITT (mITT) population (randomized and treated with at least one dose of study medication).
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 22 | 18
Participants | 3 | 2

10. Other Pre Specified Outcome: Safety TEAEs
Description: The number of subjects with treatment-emergent adverse events in each arm of all treatment-emergent adverse events (TEAEs).
Time Frame: 6 weeks
Population: Safety population includes all subjects randomized and treated with at least one dose of study medication. One subject randomized to receive placebo, was mistakenly given 2 doses of opaganib and is therefore included twice.
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 23 | 18
Participants | 11 | 9

11. Other Pre Specified Outcome: Safety SAEs
Description: The number of subjects with serious adverse events (SAEs) in each arm.
Time Frame: 6 weeks
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 23 | 18
Participants | 3 | 5

12. Post Hoc Outcome: Percent Change in Measurement of the Daily Oxygen Requirement
Description: The changes in supplemental oxygen requirement [oxygen flow (L/min)] were calculated as percent change from baseline to account for the variability of baseline values, up to Day 14. Percentage from baseline area under the (AUC) is calculated by dividing the baseline adjusted AUC with the baseline. The median AUC absolute change from baseline (L/min) for each treatment arm is presented.
Time Frame: 14 days
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Percentage of change from baseline*day
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 21 | 18
Percentage of change from baseline*day | -770.0 [-1044.3 to 0.0] | -583.6 [-916.7 to -223.3]

13. Post Hoc Outcome: Measurement of the Relative Benefit for Each Treatment Are as Derived From Oxygen Requirements
Description: The relative benefit for each treatment group derived from total oxygen requirement [area under the curve (AUC)] for each arm using daily supplemental oxygen flow (L/min) over 14 days based on the daily percent change (reduction or increase) from baseline adjusted for each subject. As the maximal possible AUC benefit of -1250% is achieved if reduction to zero (100% reduction) occurred the day after baseline and was maintained through Day 14, the relative benefit derived for each group was calculated.
Time Frame: 14 days
Population: as for outcome 2
Measure: Number; unit: Percentage of relative benefit
Arm/Group | Opaganib | Placebo
Number analyzed (Participants) | 21 | 18
Percentage of relative benefit | 61.6 | 46.7

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: One participant in the placebo arm was not dosed and therefore was removed from the safety population.
  One participant was randomized to receive placebo, was mistakenly given 2 doses of opaganib and is therefore included twice, once in each arm.
Arm/Group | Opaganib | Placebo
All-Cause Mortality (participants affected / at risk) | 3/23 | 3/18
Serious Adverse Events (participants affected / at risk) | 3/23 | 5/18
Other Adverse Events (participants affected / at risk) | 11/23 | 9/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opaganib (N=23) | Placebo (N=18)
Acute kidney injury (Renal and urinary disorders) | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opaganib (N=23) | Placebo (N=18)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Traumatic chest injury NOS (Injury, poisoning and procedural complications) | 0 | 1
Troponin I increased (Investigations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are disclosure agreements between the Sponsor and each of the participating clinical sites and PI that slightly differ.

DOCUMENTS (2):
  • Study Protocol (2020-08-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT04414618/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT04414618/SAP_001.pdf